CLINICAL TRIAL: NCT02104323
Title: Recombinant Human Endostatin Injection Study for Patients With Neurofibromatosis Type 2 (NF2) and NF2-Related Tumors by Continuous Intravenous Pumping
Brief Title: Endostatin Study for Patients With Neurofibromatosis Type 2 (NF2) and NF2-Related Tumors
Acronym: Endostatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shandong Simcere-Medgenn Bio-pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Li Peng, Li Peng, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tian-drug-neuro001; ChiCTR-ONRC-14004210 (Registry Identifier: Chinese clinical trial registry)
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Vestibular Schwannoma; Neurofibromatosis Type 2
Keywords: Neurofibromatosis Type 2; Vestibular Schwannoma; Other NF2-related tumors
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2 | interventions — Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endostatin，treatment effect evaluation (Experimental): Patients receive continuous intravenous Endostatin drug pumping during the course of treatment. The drug dosage is 7.5mg/m2/d. Every course of treatment lasts three months. Patients are designed to receive total three courses of treatment if there is no disease progression. The interval between two courses is one month.
  Interventions: Drug: Endostatin

INTERVENTIONS:
Drug: Endostatin — Method of drug administration:continuous intravenous pumping; Dosage: 7.5mg/m2/d; Course of treatment: 3 months;Total three treatment courses.
  Other Names: Recombinant Human Endostatin

SUMMARY:
1)Preliminarily evaluate the treatment effect of continuous vein injection of recombinant human endostatin on NF2; 2)Preliminarily evaluate the safety and the patient's tolerance of the treatment of endostatin; 3)Provide an objective basis for an enlarged randomized double-blind trial.

DETAILED DESCRIPTION:
Neurofibromatosis type 2 (NF2) is a hereditary tumor predisposition syndrome caused by mutations in the NF2 tumor suppressor gene. Individuals with NF2 have a higher likelihood to develop multiple nervous system tumors, including schwannomas, meningiomas, and ependymomas. The hallmark of NF2 is bilateral vestibular schwannomas. Historically, most NF2 patients experience complete hearing loss either from tumor progression or after treatment of the tumors with surgery or radiation. Effective treatments are urgently needed for NF2 patients with progressive hearing loss because hearing loss is associated with impairment in social, emotional,and communication function and with increased depression.

Previous studies of NF2 patients treated with bevacizumab suggested that inhibition of vascular endothelial growth factor (VEGF) could result in hearing improvement and reduction in tumor size.Recombinant human endostatin can inhibit the formation of blood vessels by inhibiting the migration of vascular endothelial cells .In this way, endostatin can inhibit the nutrition of the tumor and decrease the tumor's growth and metastasis. In vitro tests, endostatin can inhibit the cell migration and Tube formation of the microvascular endothelial cell line HHEC. Besides, it can inhibit blood vessels' formation of the chicken embryo sac membrane. Based on these studies, we perform this clinical trial to known the treatment effect and tolerability of endostatin on NF2.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients must be at the age of 16-30
* 2)Patients must meet the diagnostic criteria for NF2, with bilateral acoustic neuroma and other central nervous system tumors
* 3)Patients must not be treated with other drugs or radiation therapy recently
* 4)Patients should live in Beijing or nearby and can be treated in hospital
* 5)Patients must be healthy and not be seriously allergic with biological agents
* 6)Patients must join the clinical trial voluntarily, with good compliance, cooperate with the researchers well, sign a written informed consent.

Exclusion Criteria:

* 1)Treated with other drugs, surgery or radiation therapy recently
* 2)Brainstem is compressed seriously, with hydrocephalus, need to be treated with surgery in short time
* 3)Being pregnant or try to get pregnant, lactating women
* 4)With acute or chronic infectious diseases
* 5)With heart diseases, cardiac dysfunction or abnormal ECG
* 6)With uncontrolled neural or mental diseases, poor compliance
* 7)Not available for enhanced MRI
* 8)Take part in any other clinical trial
* 9)With other conditions that are considered not suitable for this clinical trial.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in volume of tumour after every course of the treatment | Baseline,Month 3,Month 7,Month 11
  Patients in this clinical trial would receive MRI test to evaluate the volume of tumour after every course of the treatment.

SECONDARY OUTCOMES:
Change from Baseline in hearing ability after every course of the treatment | Baseline,Month 3,Month 7,Month 11
  Patients' hearing ability would be tested after every course of the treatment.

OTHER OUTCOMES:
Change from baseline in QOL(quality of life) score after every course of the treatment | Baseline,Month 3,Month 7,Month 11
  Patients' QOL(quality of life) would be evaluated after every course of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pinan Liu, Study Director — Beijing Tiantan Hospital; Fu Zhao, Principal Investigator — Beijing Neurosurgical Institute
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Plotkin SR, Merker VL, Halpin C, Jennings D, McKenna MJ, Harris GJ, Barker FG 2nd. Bevacizumab for progressive vestibular schwannoma in neurofibromatosis type 2: a retrospective review of 31 patients. Otol Neurotol. 2012 Aug;33(6):1046-52. doi: 10.1097/MAO.0b013e31825e73f5. PMID 22805104
- [Background] Plotkin SR, Stemmer-Rachamimov AO, Barker FG 2nd, Halpin C, Padera TP, Tyrrell A, Sorensen AG, Jain RK, di Tomaso E. Hearing improvement after bevacizumab in patients with neurofibromatosis type 2. N Engl J Med. 2009 Jul 23;361(4):358-67. doi: 10.1056/NEJMoa0902579. Epub 2009 Jul 8. PMID 19587327
- [Background] Nunes FP, Merker VL, Jennings D, Caruso PA, di Tomaso E, Muzikansky A, Barker FG 2nd, Stemmer-Rachamimov A, Plotkin SR. Bevacizumab treatment for meningiomas in NF2: a retrospective analysis of 15 patients. PLoS One. 2013;8(3):e59941. doi: 10.1371/journal.pone.0059941. Epub 2013 Mar 21. PMID 23555840
- [Background] Plotkin SR, Ardern-Holmes SL, Barker FG 2nd, Blakeley JO, Evans DG, Ferner RE, Hadlock TA, Halpin C; REiNS International Collaboration. Hearing and facial function outcomes for neurofibromatosis 2 clinical trials. Neurology. 2013 Nov 19;81(21 Suppl 1):S25-32. doi: 10.1212/01.wnl.0000435746.02780.f6. PMID 24249803
- [Background] Mautner VF, Nguyen R, Kutta H, Fuensterer C, Bokemeyer C, Hagel C, Friedrich RE, Panse J. Bevacizumab induces regression of vestibular schwannomas in patients with neurofibromatosis type 2. Neuro Oncol. 2010 Jan;12(1):14-8. doi: 10.1093/neuonc/nop010. Epub 2009 Oct 20. PMID 20150363